CLINICAL TRIAL: NCT01935089
Title: Pilot Study: Single Arm, Multi-site, Open-label Study to Assess the Effectiveness of Peg-IFN-a2b in Decreasing the Levels of Cell-associated Integrated Viral DNA in HIV Chronic Infection
Brief Title: Pilot Peg-Interferon-a2b in Decreasing Viral DNA in HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Wistar Institute (Other)
Collaborators: University of Pennsylvania (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Luis Montaner, Professor, The Wistar Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Merck-0575
Record Dates: First submitted 2013-08-27; First posted 2013-09-04 (Estimated); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; Interferon alpha; Integrated DNA; Latent reservoir
MeSH Terms: interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interferon alpha (Experimental): pegylated Interferon alpha 2b (Pegintron) 1 µg/kg per week, 20 weeks
  Interventions: Drug: Pegylated Interferon alpha 2b

INTERVENTIONS:
Drug: Pegylated Interferon alpha 2b — 1µg/kg/week
  Other Names: Pegintron

SUMMARY:
We propose to test our primary hypothesis that treatment with Peg-IFN-α-2b will result in a decrease in integrated HIV DNA in peripheral blood and tissue in chronically HIV-infected immune-reconstituted individuals (see section 3.1) in a prospective, interventional, 1-arm, open label clinical trial. To this end, we propose to enroll 25 HIV-1-infected subjects (please refer to power calculations in section 10.1 below) currently stably suppressed (> 1y with VL < 50 copies/ml) on ART and with CD4 count > 450 cells/µl.

We hypothesize that 20 weeks of treatment with Peg-IFN-alpha-2b, in the presence of HIV reactivation (i.e.: ART interruption), will result in activation of intrinsic and/or immune-mediated anti-HIV mechanisms resulting in a decrease in the levels of viral reservoir in chronically HIV-infected, immune-reconstituted individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Body weight between 125 and 299 lbs
* Confirmed diagnosis of HIV-1 infection by western blot or by a documented HIV-1 viral load
* Currently receiving ART and on ART for > 1 year
* VL < 50 copies/ml for ≥ 1 year, with at least 2 measurements in the previous year, 1 viral "blip" with VL< 400 copies/ml allowed
* HIV viral load of <50 copies/ml at screening.
* CD4 >450 cells/µL at screening.
* A negative ECG if >45yrs men/>55yrs women years of age or if below these years of age but with two added risk factors for coronary artery disease [smoking, hypertension (BP >140/90 or on antihypertensive medications), low HDL (<40 mg/dL), family history of premature CHD (<55 yrs males/<65 females)] or a Framingham score > 15% (men) or 10% (women))

Exclusion Criteria:

* Confirmed clinical history of developing resistance to ART regimens that resulted in treatment changes
* Receiving didanosine as part of the participant's ART regimen at the time of screening
* Ongoing treatment with Isoniazide, pyrazinamide, Rifabutin, Rifampicin, Diadenosine Ganciclovir, Valgancyclovir, Oxymetholone, Thalidomide or Theophylline.
* Use of any investigational drug within 30 days prior to screening
* History or current use of immunomodulatory therapy for over 2 weeks during the 6 months prior to enrollment, including, but not limited to: IFN-alpha or gamma (recombinant or pegylated), systemic corticosteroids (nasal or pulmonary steroids will be allowed; systemic cancer chemotherapy/irradiation; cyclosporin; tacrolimus (FK-506); OKT-3; any Interleukin, including IL-2; cyclophosphamide; methotrexate; IVIG (gamma globulin); G/M-CSF; hydroxyurea; thalidomide; pentoxifylline; thymopentin; thymosin; dithiocarbonate; polyribonucleotide.
* History of adverse or allergic reactions to any type-1 interferon (e.g. IFN-alpha2a, IFN-α2b, IFN-beta)
* History of severe depression, or ongoing moderate depression determined by PHQ-9 at screening
* Type I diabetes mellitus, or type II diabetes mellitus that is not controlled with oral agents and/or insulin.
* Prior diagnosis of multiple sclerosis or other neurodegenerative disorders
* Significant co-existing lab abnormalities including:

  1. Anemia (Hgb <9.1 mg/dl men, <8.9 mg/dl women)
  2. WBC <2000 cells/µl
  3. Absolute neutrophil count (ANC) <1200 cells/ µl
  4. Platelet count <60,000 cells/ µl
  5. Liver disease (AST/ALT > 2.5x, Total Bilirubin > 1.5x upper limits of norm (ULN), or Total Bilirubin >3x ULN if receiving indinavir OR Atazanavir)
  6. Renal disease (creatinine > 2x upper normal limits or creatinine clearance <60mg/dl (by Crockoff-Gault)
* Chronic HCV infection (HCV viremia), or HBV Ag positive and/ or HBV viremia (Notice: subjects with prior HCV infection with a documented sustained virologic response with treatment finishing >1 year prior to screening are eligible for enrollment).
* Liver cirrhosis or hepatic decompensation with Child Pugh score > 6
* History of major organ transplantation with an existing functional graft.
* Evidence of OI or other active infectious diseases or active malignancies
* Active Autoimmune diseases, including autoimmune hepatitis
* History of retinopathy or clinically significant ophthalmologic disease on eye exam performed within 6 months prior to initiation of IFN
* Pregnancy, actively attempting to become pregnant, or breastfeeding
* Body weight under 125 lbs or over 300 lbs
* Other conditions, such as active drug/alcohol abuse or dependence which would interfere with study compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08-07; Primary Completion 2015-03-25 (Actual); Study Completion 2016-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis J Montaner, DPhil, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - AIDS Clinical Trials Unit (ACTU), and Department of Medicine, University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Presbyterian Hospital, Department of Medicine, University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Jonathan Lax Clinic, Philadelphia FIGHT, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Papasavvas E, Azzoni L, Ross BN, Fair M, Howell BJ, Hazuda DJ, Mounzer K, Kostman JR, Tebas P, Montaner LJ. Comparable HIV suppression by pegylated-IFN-alpha2a or pegylated-IFN-alpha2b during a 4-week analytical treatment interruption. AIDS. 2021 Oct 1;35(12):2051-2054. doi: 10.1097/QAD.0000000000002961. PMID 34049356
- [Derived] Papasavvas E, Azzoni L, Pagliuzza A, Abdel-Mohsen M, Ross BN, Fair M, Howell BJ, Hazuda DJ, Chomont N, Li Q, Mounzer K, Kostman JR, Tebas P, Montaner LJ. Safety, Immune, and Antiviral Effects of Pegylated Interferon Alpha 2b Administration in Antiretroviral Therapy-Suppressed Individuals: Results of Pilot Clinical Trial. AIDS Res Hum Retroviruses. 2021 Jun;37(6):433-443. doi: 10.1089/AID.2020.0243. Epub 2021 Jan 29. PMID 33323024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 screened
Period: Overall Study
Arm/Group | Interferon Alpha
Started | 20
Completed | 17
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Interferon Alpha
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [40.5 to 53.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
CD4 count [Median (Inter-Quartile Range); unit: cells/ul] | 591 [545.25 to 906.5]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Copies of HIV DNA Per CD4+ T Cell at Week 24
Description: Difference in copies of HIV DNA per CD4+ T cell between baseline and week 24, assessed by Alu-HIVgag polymerase chain reaction
Time Frame: Week 3 and 24
Population: outcome measure available only for 17 individuals
Measure: Median (Inter-Quartile Range); unit: HIV DNA copies per CD4+ T cell
Arm/Group | Interferon Alpha
Number analyzed (Participants) | 17
HIV DNA copies per CD4+ T cell
  Baseline | 113 [65 to 371]
  Week 24 | 98 [60 to 406.5]
Statistical Analysis 1: Comparison: Interferon Alpha; Test type: Other — Hypothesis: 20 weeks of treatment (baseline week 3 to endpoint week 24) will result in a change in the levels of integrated HIV-1 DNA (copies/CD4 T cell Variable name: intDNA). Test if the mean difference (IntDNA wk24 - IntDNAwk3) is significantly different from zero (i.e. no change) Null hypothesis: Mean (IntDNA wk24 - IntDNAwk3) = 0; reject if p<0.05; p = 0.0797, signed rank test — significant if <0.05

ADVERSE EVENTS:
Arm/Group | Interferon Alpha
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 11/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Alpha (N=20)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) — grade 4 neutropenia requiring treatment discontinuation. Not SUSAR
Neutropenia (Blood and lymphatic system disorders) | 6 (6) — Lower grade neutropenia managed with treatment or dose reduction
Depression (Nervous system disorders) | 3 (3) — grade 2 depression managed with medication. One individual chose to withdraw from study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes